CLINICAL TRIAL: NCT01801501
Title: Role of FGF-23 as a Prognosis Biomarker in Intensive Care Patients
Status: Completed | Type: Observational
Sponsor: University of Chile (Other)
Responsible Party: Principal Investigator, Luis Toro, Physician, University of Chile
Other Study IDs: AKI-FGF23-012
Record Dates: First submitted 2013-02-25; First posted 2013-02-28 (Estimated); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Sepsis; Acute Kidney Injury
MeSH Terms: conditions — Sepsis; Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: Samples Without DNA — Venous blood samples will be obtained. Serum samples will be extracted, with elimination of other material. Serum will be stored at -20ºC until plasma molecules determination was performed by ELISA technique.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Critical Care Patients: Patients admitted in Critical Care Unit with diagnosis of severe sepsis/septic shock

SUMMARY:
The purpose of the study is to evaluate the potential role of plasmatic Fibroblast Growth Factor 23 (FGF-23) as a prognosis predictor of clinical outcomes in Critical Care patients.

DETAILED DESCRIPTION:
Observational study of patients admitted in the Critical Care Unit (CCU) of University of Chile Clinical Hospital, admitted with diagnosis of severe sepsis/septic shock.

Exclusion criteria: Pregnancy, organ transplantation. Informed consent is solicited to patients before admission in study. If the patient cannot give it because of his/her clinical condition, it will be solicited to a patient representative.

After admission in CCU and achievement of informed consent, a venous blood sample will be obtained, to determinate plasmatic levels of Fibroblast Growth Factor 23 (FGF-23). New samples will be obtained at 24 and 48 hours after admission. Determination of FGF-23 will be performed by ELISA technique in Integrated Physiology laboratory.

Demographics, clinical and biochemical data will also be obtained. The data will be collected by the Principal Investigator. Confidentially of all data will be preserved during and after the completion of the study.

The study is divided in 2 parts:

1. - Evaluation of a sample of 14 patients to determinate the impact of FGF-23 to predict presence and severity of Acute Kidney Injury (AKI), and to estimate sample size to predict primary outcomes.
2. - Evaluation of a larger sample, to determinate the impact of FGF-23 to predict primary outcomes.

Primary outcomes:

1. - Development of acute kidney injury
2. - Severity of AKI, determinate by AKIN classification
3. - In-hospital mortality

Secondary outcomes:

1. - Requirements of renal replacement therapy
2. - Requirements of mechanical ventilation
3. - Requirements of vasoactive drugs
4. - Duration of ICU stay and hospital stay

As a post-hoc analysis, we performed a measurement of a combined biomarker, including FGF-23 and other 2 biomarkers, Klotho and Erythropoietin, measured in blood samples, to determinate its predictive capacity for AKI diagnosis and mortality.

The protocol was approved by the Ethical Committee of University of Chile Clinical Hospital. The study is monitored by the Clinical Investigation Support Office (OAIC) of the hospital.

ELIGIBILITY:
Inclusion Criteria:

* Admission in Critical Care Unit
* Sepsis

Exclusion Criteria:

* Pregnancy
* Organ transplantation

Ages: 15 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients admitted in Critical Care Unit with diagnosis of severe sepsis/septic shock.
  Pregnant women and transplanted patients are excluded.
Sampling Method: Probability Sample
Enrollment: 164 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2014-04 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Overall survival | 30 days and 1 year
  Determination of overall survival during the first 30 days and 1 year after admission

SECONDARY OUTCOMES:
Duration of hospitalization | 30 days
  Determination of number of days of hospitalization (in ICU and overall hospitalization)

OTHER OUTCOMES:
Development of acute kidney injury | 30 days
  Evaluation of development of AKI, using KDIGO creatinine criteria

CONTACTS AND LOCATIONS:
Overall Officials: Luis Toro, MD, Principal Investigator — University of Chile Clinical Hospital; Luis Michea, MD PhD, Principal Investigator — University of Chile; Carlos Romero, MD, Study Chair — University of Chile Clinical Hospital
Locations (1):
- University of Chile Clinical Hospital, Santiago, RM, Chile